CLINICAL TRIAL: NCT01764711
Title: Aldosterone and Sodium Regulation in Postural Tachycardia Syndrome Aim 1b: ACTH Stimulation
Brief Title: Adrenocorticotropic Hormone Stimulation in Postural Orthostatic Tachycardia Syndrome (POTS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alfredo Gamboa, Research Associate Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 121548; R01HL102387 (NIH)
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Postural Tachycardia Syndrome
Keywords: POTS
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Cosyntropin

ARMS (2):
- Low Salt Diet POTS (Experimental): Each participant will be asked to sit in a chair for 30 minutes prior to a blood draw. Then a small dose of cosyntropin is administered intravenous. Blood samples will be drawn again at 30 minutes and 60 minutes after the drug has been given.
  Interventions: Drug: Cosyntropin administration
- Low Sodium Diet Controls (Experimental): Each participant will be asked to sit in a chair for 30 minutes prior to a blood draw. Then a small dose of cosyntropin is administered intravenous. Blood samples will be drawn again at 30 minutes and 60 minutes after the drug has been given.
  Interventions: Drug: Cosyntropin administration

INTERVENTIONS:
Drug: Cosyntropin administration — After 30 minutes of rest in the seated position, participants will be given cosyntropin intravenously. Blood samples will be taken 30 minutes pre-drug administration, 30 minutes post and 60 minutes post drug administration.
  Other Names: Cortrosyn

SUMMARY:
This study is to determine different chemical levels in the blood during a low salt diet. This study will compare normal volunteers to those with Postural Tachycardia Syndrome (POTS)

DETAILED DESCRIPTION:
Patients with postural tachycardia syndrome had a subnormal increment in aldosterone with upright posture, which might reflect a blunted adrenal response to stimulation upon assuming upright posture. In this AIM, we propose to assess the adrenal response to aldosterone stimulation with intravenous adrenocorticotropin hormone.

For this protocol, subjects enrolled in the parent study will be approached about this sub-study. Subjects will be assured that they are not required to participate in this study even if they choose to participate in the parent study.

There will be no randomization for this specific sub-study. The order of diets (low sodium vs. high sodium) will be performed as a part of the parent study, and not as a part of this sub-study. This sub-study will only be performed in the LOW dietary salt phase.

All subjects will be previously screened and evaluated as a part of the parent study. No further screening will be performed exclusively for this study. Women of childbearing potential will have had a serum pregnancy test as a part of the parent study. Pregnant women will not be allowed to participate.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be enrolled in the parent study "Dietary Salt in Postural Tachycardia Syndrome" during the "LOW SALT" phase

Postural Tachycardia Syndrome Diagnosed with postural tachycardia syndrome by the Vanderbilt Autonomic Dysfunction Center Increase in heart rate ≥30 beats/min with position change from supine to standing (10 minutes) Chronic symptoms consistent with POTS that are worse when upright and get better with recumbence

* Control Subjects

  * Healthy, non-obese, non-smokers without orthostatic tachycardia
  * Selected to match profiles of POTS patients (gender, age)
  * Not using vasoactive medication
* Age between 18-50 years
* Male and female subjects are eligible.
* Able and willing to provide informed consent

Exclusion Criteria:

* Overt cause for postural tachycardia (such as acute dehydration)
* Inability to give, or withdrawal of, informed consent
* pregnant
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2013-01; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo J Gamboa, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Salt Diet Controls: Each participant will be asked to sit in a chair for 30 minutes prior to a blood draw. Then a small dose of cosyntropin is administered intravenous. Blood samples will be drawn again at 30 minutes and 60 minutes after the drug has been given.
  Cosyntropin administration: After 30 minutes of rest in the seated position, participants will be given cosyntropin intravenously. Blood samples will be taken 30 minutes pre-drug administration, 30 minutes post and 60 minutes post drug administration.
Period: Overall Study
Arm/Group | Low Salt Diet POTS | Low Salt Diet Controls
Started | 8 | 5
Completed | 8 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Salt Diet POTS; Low Salt Diet Controls: After 7 days of being on a low salt diets, POTS patients and controls will be asked to undergo Cosyntropin administration: After 30 minutes of rest in the seated position, participants will be given cosyntropin intravenously. Blood samples will be taken 30 minutes pre-drug administration, 30 minutes post and 60 minutes post drug administration.
- Total: Total of all reporting groups
Arm/Group | Low Salt Diet POTS | Low Salt Diet Controls | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (6) | 30 (8) | 32 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 13
Baseline Aldosterone [Mean (Standard Deviation); unit: nanograms/dL] | 34 (20.1) | 33 (14.2) | 33.5 (16.2)

OUTCOME MEASURES:

1. Primary Outcome: Alldosterone Increase in Response to Adrenocorticotropin Hormone (ACTH).
Description: To assess the adrenal responsiveness to adrenocorticotropin hormone (ACTH), as measured by plasma aldosterone level, is contributing to the pathophysiology of Orthostatic Tachycardia.
Time Frame: 30 minutes after injection of ACTH
Measure: Mean (Standard Deviation); unit: nanograms/dL
Arm/Group | Low Salt Diet POTS | Low Salt Diet Controls
Number analyzed (Participants) | 8 | 5
nanograms/dL | 52.5 (15.7) | 57.9 (26.4)

ADVERSE EVENTS:
Time Frame: Adverse events were assess for two hours after administration of ACTH.
Arm/Group | Low Salt Diet POTS | Low Salt Diet Controls
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 0/8 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-07-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT01764711/Prot_SAP_ICF_000.pdf